CLINICAL TRIAL: NCT02823431
Title: Contribution of Urethral Sensory Feedback in Voiding Efficiency
Brief Title: Effect of Urethral Analgesia on Voiding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00071589
Record Dates: First submitted 2016-04-28; First posted 2016-07-06 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2017-10

CONDITIONS: Urethral Analgesia
Keywords: voiding efficiency; detrusor underactivity; urodynamics
MeSH Terms: conditions — Urinary Bladder, Underactive | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Analgesia Arm (Active Comparator): Participants randomized to this arm will undergo uroflow studies then be given a 2-hour rest. Urodynamics with the use of Urojet (lidocaine hydrochloride 2%) will then be performed. The lidocaine gel will be placed in and around the urethra. It will be allowed to set for 3 minutes, then the remainder of the standard urodynamic evaluation will be performed. We are using Urojet (lidocaine gel) in an FDA approved manner (for analgesia).
  Interventions: Drug: lidocaine gel
- Placebo Arm (Placebo Comparator): Participants randomized to this arm will first undergo uroflow studies then be given a 2-hour rest. Urodynamic testing without analgesia (standard of care) will then be performed.
  Interventions: Other: Plain aqueous gel

INTERVENTIONS:
Drug: lidocaine gel
  Other Names: Urojet 2% gel
  Arms: Analgesia Arm
Other: Plain aqueous gel
  Other Names: KY gel
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to evaluate how urethral analgesia impacts voiding efficiency in healthy women. The investigator hypothesizes that anesthetizing the urethral with lidocaine gel will decrease voiding efficiency as measured by standard bladder testing (urodynamic testing).

DETAILED DESCRIPTION:
1. Purpose of the Study The purpose of this study is to determine whether urethral sensory feedback has a role in the micturition (bladder emptying) reflex in female controls during routine office Urodynamic Studies (UDS). UDS are current clinical tests of urethral and bladder function and consist of several individual studies including filling cystometry, pressure-flow studies, and urethral pressure profilometry (UPP). Filling cystometry focuses primarily on sensation and activity of the bladder during the filling (or storage) phase of the micturition (voiding) cycle. Pressure-flow studies (which include voiding cystometry) are used to assess the motor activity of the bladder muscle during bladder emptying. UPP assesses urethral sphincter motor function and has traditionally been used to evaluate stress urinary incontinence. Perineal patch electromyography (EMG) is often added to UDS to assess for pelvic floor muscle recruitment during voiding, which may suggest voiding dysfunction.
2. Background & Significance The storage and elimination of urine is regulated by neural circuits in the brain and spinal cord to coordinate function between the urinary bladder and the urethra. During the micturition (bladder emptying) reflex, the elimination of urine is facilitated by bladder wall contraction and urethral wall and pelvic floor muscle relaxation. Urine that subsequently flows through the urethra also activates sensory nerves to amplify bladder contractions and maintain efficient bladder emptying. Incomplete voiding and urinary retention occurs when these mechanisms are disrupted or poorly coordinated.

   Incomplete bladder emptying due to detrusor underactivity is an understudied health concern for women in the United States. The overall incidence detrusor underactivity in women has not yet been reported in the literature. One study by Wu et al. (2005) determined that 7.8% of patients in an outpatient rehabilitation facility had symptoms of incomplete bladder emptying; whereas, 21% of people without symptoms had elevated post void residuals when universally screened. Their population consisted of 350 patients, of which two-thirds were women. Lower urinary tract symptoms, including urinary urgency, frequency and incomplete bladder emptying, have been shown to decrease quality of life, increase healthcare utilization, decrease workplace productivity, and impact intimate relationships.

   The current clinical management options for women with retention are intermittent or indwelling catheterization, urethral dilation, or reconstructive surgery. These treatments, however, often fail to completely resolve lower urinary tract symptoms and the patients may develop chronic retention complications such as overflow incontinence, hydroureter, hydronephrosis, infection, or renal failure. In order to improve therapeutic outcomes, there is still a need to clarify the specific mechanisms that underlie detrusor underactivity in women. Our proposed studies will be contributing to the growing body of literature implicating urethral sensory feedback as a candidate to recover efficient bladder emptying.
3. Hypothesis and Justification Overall Hypothesis: Urethral afferent nerve fiber activation augments bladder contractions for efficient voiding and urethral anesthesia will disrupt sensory feedback and impair bladder emptying.

   Specific Aim 1: To assess voiding efficiency (voided volume/{voided volume + residual volume}) in women controls with and without urethral anesthesia Hypothesis 1a: Voiding efficiency will be lower when the urethra is anesthetized during micturition pressure-flow studies Hypothesis 1b: Detrusor contraction at maximum flow rate (Pdet@Qmax) and duration of detrusor contraction will be reduced when the urethra is anesthetized during micturition pressure-flow studies Hypothesis 1c: Voiding while anesthetized will lead to increased valsalva-voiding (increased intra-abdominal pressure, Pabd) and an intermittent urinary stream during micturition pressure-flow studies

   Specific Aim 2: To assess whether urethral anesthesia gel improves discomfort during the UDS Hypothesis: Visual Analog Scale (VAS) scores for pain will be lower during the UDS when the urethra has been anesthetized

   Studies supporting Specific Aims:

   i. Micturition with Urethral Anesthesia Distension and fluid flow in the urethra has been previously demonstrated to evoke sensory nerve discharge. Nerve firing originating from the urethra is then able to initiate contractions in the filling bladder and increase the amplitude and duration of ongoing bladder contractions. This pudendal-bladder reflex has been shown to be necessary for efficient bladder emptying because disruption to urethral sensory feedback by transection of the sensory branch of the pudendal nerve or intraurethral anesthesia reduces voiding efficiency in the rat. Urethral anesthesia in humans has also been demonstrated to increase post void residual and alter symptoms experienced during the voiding phase.

   This investigator's approach is novel as this study will characterize voiding in healthy women who will be randomized to placebo versus urethral analgesia. Investigators will do this by performing UDS, which will include all clinical tests for bladder function, with or without urethral anesthesia (2% lidocaine hydrochloride jelly or plain aqueous gel).

   ii. Pain Perception During Catheterization Urethral catheterization elicits mild to moderate pain in women. The use of lubricant anesthetic on the catheter is one available option to manage tissue trauma and pain perception. Several studies have reported that 2% lidocaine gel reduces procedural pain during female urethral catheterization. Others however, have found that lubricant anesthetic and catheter size, does not effect the perception of pain in urethral catheterization in women. These discrepant reports suggest a consensus has not been reached on the efficacy of lubricant anesthetic and pain perception in women.
4. Subject Recruitment: Subjects will be recruited from Duke Hospital and Duke University Campus via newspaper advertisements and paper fliers.
5. Design and Procedures To account for screen failures, it is anticipated that a total of 40 female controls will be screened to achieve n=20 for completed UDS. Subjects will perform a baseline voiding test (uroflow), then will be randomized to undergoing urodynamic studies with or without urethral analgesia. Participants will be randomized to their arm of the study using a random number generator (MatLab). Study staff and the subjects will be blinded to the treatment regimen; thus, this study design is a randomized double-blind placebo-controlled trial. Inclusion and exclusion criteria are listed in a separate section.

Study Visit Questionnaires and Tests After their phone screen, (3.i), participants will be scheduled for the study visit. All study procedures will take place at the Duke Urogynecology Office at Patterson Place. Participants will undergo informed consent on arrival to their study visit. Subjects will provide a urine specimen for a point of care urinalysis and pregnancy test. Pre-procedure vital signs, including height and weight will be obtained. Subjects will fill out the following questionnaires: Lower Urinary Tract Symptoms Tool, Sociodemographics and Functional Comorbidity Index and complete a Medication List.

If subjects have a negative urinalysis and pregnancy test they will be randomized. If either of their point of care tests is positive (per exclusion criteria), they will be excluded from the study and referred to their primary care physician.

Prior to performing UDS, the subject's bladder will be scanned transabdominally with a standard clinic bladder scanner. This will ensure adequate urine is within the bladder to start the first test.

The participant will then be placed in the dorsal lithotomy position and a pelvic exam will be performed to confirm no pelvic organ prolapse past the hymen during valsalva. Uroflow testing will then begin. Subjects will then undergo a 2-hour wait and be given water to re-fill their bladder. After two hours, Urodynamic testing will be performed.

Order of Studies Performed During Urodynamic Testing: Complex Uroflowmetry, Complex Cystometry, Urethral Pressure Profilometry, Micturition Pressure-flow Study

The Visual Analog Scale (VAS) will be administered to assess discomfort at the following times; after uroflow but before PVR (baseline), immediately after the urethral catheter is placed, after 100mL of fluid has been instilled, and at full bladder capacity (MCC).

After the completion of the UDS procedures, subjects will have completed their study visit.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18-60 years
* No health conditions as indicated in exclusion criteria
* Able to provide informed consent and agree to the risks of the study
* Willing to abstain from caffeine and alcohol for 24 hours
* Willing to avoid taking anticholinergic medications (for reasons other than incontinence; e.g., diphenhydramine) for one week prior to the procedure

Exclusion Criteria:

* Pelvic organ prolapse past the hymen
* Multiple sclerosis, myasthenia gravis, Parkinson's Disease, stroke within the past 6 months
* Interstitial cystitis / Bladder Pain Syndrome
* Recurrent (≥ 3/year) urinary tract infections
* Positive pregnancy test at the time of consent
* ≤ 6 weeks postpartum or if breastfeeding
* Positive urine dip (>+1nitrites or >1+LE) and urinary symptoms at the time of consent
* >1+ blood on urinary dip
* Morbid obesity (BMI >40)
* Taking anticholinergic medications for urinary incontinence
* >2 replies of ≥ "sometimes" on the Lower Urinary Tract Symptoms questionnaire at the time of consent

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren Grill, Principal Investigator — Duke University
Locations (1):
- Duke University Campus, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SC, Grill WM, Fan WJ, Kou YR, Lin YS, Lai CH, Peng CW. Bilateral pudendal afferent stimulation improves bladder emptying in rats with urinary retention. BJU Int. 2012 Apr;109(7):1051-8. doi: 10.1111/j.1464-410X.2011.10526.x. Epub 2011 Aug 23. PMID 21883860
- [Background] Peng CW, Chen JJ, Cheng CL, Grill WM. Improved bladder emptying in urinary retention by electrical stimulation of pudendal afferents. J Neural Eng. 2008 Jun;5(2):144-54. doi: 10.1088/1741-2560/5/2/005. Epub 2008 Apr 22. PMID 18430976
- [Background] Shafik A, Shafik AA, El-Sibai O, Ahmed I. Role of positive urethrovesical feedback in vesical evacuation. The concept of a second micturition reflex: the urethrovesical reflex. World J Urol. 2003 Aug;21(3):167-70. doi: 10.1007/s00345-003-0340-5. Epub 2003 Jul 25. PMID 12898170
- [Derived] Kisby CK, Gonzalez EJ, Visco AG, Amundsen CL, Grill WM. Randomized Controlled Trial to Assess the Impact of Intraurethral Lidocaine on Urodynamic Voiding Parameters. Female Pelvic Med Reconstr Surg. 2019 Jul/Aug;25(4):265-270. doi: 10.1097/SPV.0000000000000544. PMID 29300256

RESULTS

PARTICIPANT FLOW:
Groups:
- Analgesia Arm: Participants randomized to this arm will undergo uroflow studies then be given a 2-hour rest. Urodynamics with the use of Urojet (lidocaine hydrochloride 2%) will then be performed. The lidocaine gel will be placed in and around the urethra. It will be allowed to set for 3 minutes, then the remainder of the standard urodynamic evaluation will be performed. We are using Urojet (lidocaine gel) in an FDA approved manner (for analgesia).
  lidocaine gel
- Placebo Arm: Participants randomized to this arm will first undergo uroflow studies then be given a 2-hour rest. Urodynamic testing without analgesia (standard of care) will then be performed.
  Plain aqueous gel
Period: Overall Study
Arm/Group | Analgesia Arm | Placebo Arm
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Analgesia Arm | Placebo Arm | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (9.6) | 33 (9.2) | 31.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23 (3.7) | 25 (5) | 24 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Voiding Efficiency
Description: voided volume/{voided volume + residual volume} during micturition study during urodynamic studies
Time Frame: duration of urodynamic study, 2 hours
Measure: Mean (Standard Deviation); unit: Percent voiding efficiency
Arm/Group | Analgesia Arm | Placebo Arm
Number analyzed (Participants) | 11 | 12
Percent voiding efficiency | 87 (8) | 90 (5)

2. Secondary Outcome: Detrusor Pressure at Maximum Flow
Description: bladder pressure reading (mmHg) during maximum flow during micturition
Time Frame: duration of urodynamic study, 2 hours
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Analgesia Arm | Placebo Arm
Number analyzed (Participants) | 11 | 12
cmH2O | 37.6 (19.2) | 31 (18.9)

3. Secondary Outcome: Number of Participants With Interrupted Urinary Flow Pattern During Micturition
Description: presence of interrupted flow during micturition
Time Frame: duration of urodynamic study, 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Analgesia Arm | Placebo Arm
Number analyzed (Participants) | 11 | 12
Participants | 4 | 0

4. Secondary Outcome: Visual Analog Scale Scores (Measure of Discomfort) After Catheterization
Description: visual analog scales were performed to evaluate discomfort at specified time points during the urodynamic studies. The scale is 1-100mm, with higher numbers indicating greater discomfort.
Time Frame: duration of urodynamic study, 2 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Analgesia Arm | Placebo Arm
Number analyzed (Participants) | 11 | 12
mm | 26 (20) | 19 (21)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study visit and if contact was made by the participant in the 1 month following the study visit.
Arm/Group | Analgesia Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No